CLINICAL TRIAL: NCT04967937
Title: Neuromuscular Training Improves Single-Limb Stability in Young Female Athletes
Brief Title: Neuromuscular Training Improves Single-Limb Stability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REC/Lhr/21/0414 Shah bano
Record Dates: First submitted 2021-07-19; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: ACL Injury
Keywords: Single limb stability; Neuromuscular Training; Female athletes; ACL
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-Group (Experimental): The neuromuscular training program will consist of three 90-minute training sessions per week for 6 weeks. The 3 components of the dynamic neuromuscular training protocol utilized in this study include: (1) balance training and hip/pelvis/trunk strengthening, (2) plyometrics and dynamic movement training, and (3) resistance training. Following the completion of the training program, each subject will be re-evaluated to determine change in total, anterior-posterior, and medial-lateral single-limb stability. Two-way analysis of variance models will be used to determine differences between pre-training and post-training and between limbs.
  Interventions: Other: Strengthening, resistance exercise, plyometric and dynamic movement training

INTERVENTIONS:
Other: Strengthening, resistance exercise, plyometric and dynamic movement training — (1) balance training and hip/pelvis/trunk strengthening, (2) plyometrics and dynamic movement training, and (3) resistance training.

SUMMARY:
Pretest/post-test study design, study will try to determine if a 6-week neuromuscular training program designed to decrease the incidence of anterior cruciate ligament (ACL) injuries would improve single-limb stability in young female athletes. Healthy female high school athletes will participate in this study. Single-limb postural stability for both lower extremities will be assessed with Stork balance test, Star Excursion Balance Test for Dynamic Balance and Single leg stance test for static balance. Participants will be included through convenient sampling. Informed consent will be taken from all the participants.

DETAILED DESCRIPTION:
In this Controlled single-group pretest/post-test study design, study will try to determine if a 6-week neuromuscular training program designed to decrease the incidence of anterior cruciate ligament (ACL) injuries would improve single-limb stability in young female athletes. Current study hypothesized that neuromuscular training would result in an improvement of postural stability, with the greatest improvement taking place in the medial-lateral direction. Healthy female high school athletes will participate in this study. Single-limb postural stability for both lower extremities will be assessed with Stork balance test, Star Excursion Balance Test for Dynamic Balance and Single leg stance test for static balance. Participants will be included through convenient sampling. Informed consent will be taken from all the participants. Those individuals who will match the inclusion and exclusion criteria will be a part of the study. The neuromuscular training program will consist of three 90-minute training sessions per week for 6 weeks. Following the completion of the training program, each subject will be re-evaluated to determine change in total, anterior-posterior, and medial-lateral single-limb stability.

ELIGIBILITY:
Inclusion Criteria:

* Age will range from 13-20
* Female participants
* Individuals with Postural instability and Impaired balance will be included.

Exclusion Criteria:

* Any malignancy
* Infection
* Systemic illness
* Trauma

Ages: 13 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Female athletes
Enrollment: 20 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
i. Star Excursion Balance Test for Dynamic Balance | 6th Week
  dynamic test that requires strength, flexibility, and proprioception. It is a measure of dynamic balance that provides a significant challenge to athletes and physically active individuals. The test can be used to assess physical performance

SECONDARY OUTCOMES:
ii. Single Limb Stance Test (Static Posture and Balance) | 6th Week
  The Single leg Stance (SLS) Test is used to assess static postural and balance control.Performed with eyes open and hands on the hips.Client must stand unassisted on one leg

OTHER OUTCOMES:
iii. Stork balance test | 6th Week
  The standing stork test monitors the progress of the athletes' abilities to maintain balance in a static position. This test monitors the balance of athletes because the more balance you have as an athlete, the better you may perform on the field and the fewer injuries you are likely to sustain.

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil Ur Rehman, Principal Investigator — Riphah International University
Locations (1):
- Samnabad Sports complex, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Etty Griffin LY. Neuromuscular training and injury prevention in sports. Clin Orthop Relat Res. 2003 Apr;(409):53-60. doi: 10.1097/01.blo.0000057788.10364.aa. PMID 12671485
- [Background] Richmond SA, Kang J, Doyle-Baker PK, Nettel-Aguirre A, Emery CA. A School-Based Injury Prevention Program to Reduce Sport Injury Risk and Improve Healthy Outcomes in Youth: A Pilot Cluster-Randomized Controlled Trial. Clin J Sport Med. 2016 Jul;26(4):291-8. doi: 10.1097/JSM.0000000000000261. PMID 27367045
- [Background] McLeod TC, Armstrong T, Miller M, Sauers JL. Balance improvements in female high school basketball players after a 6-week neuromuscular-training program. J Sport Rehabil. 2009 Nov;18(4):465-81. doi: 10.1123/jsr.18.4.465. PMID 20108849
- [Background] Gianotti SM, Marshall SW, Hume PA, Bunt L. Incidence of anterior cruciate ligament injury and other knee ligament injuries: a national population-based study. J Sci Med Sport. 2009 Nov;12(6):622-7. doi: 10.1016/j.jsams.2008.07.005. Epub 2008 Oct 2. PMID 18835221
- [Background] Viola RW, Steadman JR, Mair SD, Briggs KK, Sterett WI. Anterior cruciate ligament injury incidence among male and female professional alpine skiers. Am J Sports Med. 1999 Nov-Dec;27(6):792-5. doi: 10.1177/03635465990270061701. PMID 10569367
- [Background] Bonci CM. Assessment and evaluation of predisposing factors to anterior cruciate ligament injury. J Athl Train. 1999 Apr;34(2):155-64. PMID 16558559
- [Background] Hewett TE, Lindenfeld TN, Riccobene JV, Noyes FR. The effect of neuromuscular training on the incidence of knee injury in female athletes. A prospective study. Am J Sports Med. 1999 Nov-Dec;27(6):699-706. doi: 10.1177/03635465990270060301. PMID 10569353
- [Background] Myer GD, Ford KR, Brent JL, Hewett TE. Differential neuromuscular training effects on ACL injury risk factors in"high-risk" versus "low-risk" athletes. BMC Musculoskelet Disord. 2007 May 8;8:39. doi: 10.1186/1471-2474-8-39. PMID 17488502
- [Background] Chappell JD, Limpisvasti O. Effect of a neuromuscular training program on the kinetics and kinematics of jumping tasks. Am J Sports Med. 2008 Jun;36(6):1081-6. doi: 10.1177/0363546508314425. Epub 2008 Mar 21. PMID 18359820
- [Background] Hewett TE, Ford KR, Myer GD. Anterior cruciate ligament injuries in female athletes: Part 2, a meta-analysis of neuromuscular interventions aimed at injury prevention. Am J Sports Med. 2006 Mar;34(3):490-8. doi: 10.1177/0363546505282619. Epub 2005 Dec 28. PMID 16382007
- [Background] Ireland ML. Anterior cruciate ligament injury in female athletes: epidemiology. J Athl Train. 1999 Apr;34(2):150-4. PMID 16558558
- [Background] Myer GD, Sugimoto D, Thomas S, Hewett TE. The influence of age on the effectiveness of neuromuscular training to reduce anterior cruciate ligament injury in female athletes: a meta-analysis. Am J Sports Med. 2013 Jan;41(1):203-15. doi: 10.1177/0363546512460637. Epub 2012 Oct 9. PMID 23048042